CLINICAL TRIAL: NCT01029860
Title: A Study Investigating the Impact of Hospitalization on Ambulatory Blood Pressure and Intraocular Pressure in Subjects With Mild to Moderate Arterial Hypertension and Untreated Ocular Hypertension
Brief Title: The Impact of Hospitalization on Ambulatory Blood Pressure and Intraocular Pressure
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Anastasios Lasaridis, 1st Department of Internal Medicine, Aristotle University, Thessaloniki
Other Study IDs: A3244
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2007-03

CONDITIONS: Blood Pressure
Keywords: Hypertension; Ambulatory measurement
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the effect of hospital admission on 24-hour ambulatory blood pressure (ABP) in hypertensive subjects.Treated or untreated hypertensive adults with open angle glaucoma underwent in-hospital and outpatient 24-hour ABP monitoring, in random order 4 weeks apart.

ELIGIBILITY:
Inclusion Criteria:

* age >30 years old.
* subject has signed an informed consent.
* patient has untreated ocular hypertension (IOP at 10:00 between 22-34 mm Hg)
* patient has stage 1 arterial hypertension with or without therapy

Exclusion Criteria:

* secondary hypertension.
* stage 2 or 3 hypertension, history of renal disease.
* sleep apnea.
* diabetes mellitus
* acute or chronic inflammation.
* myocardial infarction or unstable angina within the past 6 months.
* heart failure NYHA class III-IV.
* active liver disease.
* pregnancy.
* history of drug or alcohol abuse, or any other condition with poor prognosis.
* treatment with non-steroid anti-inflammatory agents, corticosteroids, beta-blockers, or any other regimen that could affect BP levels.
* smoking

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with untreated ocular hypertension and stage 1 arterial hypertension with or without treatment with anti-hypertensive agents.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)